CLINICAL TRIAL: NCT01939275
Title: 64Cu-DOTA-trastuzumab Positron Emission Tomography in Patients With Gastric Cancer
Brief Title: 64Cu DOTA-Trastuzumab PET/CT in Studying Patients With Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13229; NCI-2013-01721 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13229 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage IA Gastric Cancer; Stage IB Gastric Cancer; Stage IIA Gastric Cancer; Stage IIB Gastric Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — 64Cu-DOTA-trastuzumab; Positron-Emission Tomography; Tomography, Emission-Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (copper Cu 64-DOTA-trastuzumab PET scan) (Experimental): Patients receive copper Cu 64-DOTA-trastuzumab IV on day 1 and then undergo PET/CT scan on days 2 or 3.
  Interventions: Radiation: copper Cu 64-DOTA-trastuzumab; Device: positron emission tomography; Other: laboratory biomarker analysis; Procedure: Computed Tomography

INTERVENTIONS:
Radiation: copper Cu 64-DOTA-trastuzumab — Undergo Copper Cu 64-DOTA-trastuzumab PET/CT scan
  Other Names: 64Cu-DOTA-trastuzumab
Device: positron emission tomography — Undergo Copper Cu 64-DOTA-trastuzumab PET/CT scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: laboratory biomarker analysis — Correlative studies
Procedure: Computed Tomography — Undergo Copper Cu 64-DOTA-trastuzumab PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography

SUMMARY:
This pilot clinical trial studies copper Cu 64 (64Cu) tetra-azacyclododecanetetra-acetic acid (DOTA)-trastuzumab positron emission tomography (PET)/computed tomography (CT) in studying patients with gastric, or stomach cancer. Diagnostic procedures, such as copper Cu 64-DOTA-trastuzumab PET/CT, may help doctors study the characteristics of tumors and choose the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare tumor uptake of 64Cu-DOTA-trastuzumab (copper Cu 64-DOTA-trastuzumab) in gastric cancer patients with pathologic evaluation of tumor human epidermal growth factor receptor 2 (HER2)/neu expression.

II. To compare copper Cu 64-DOTA-trastuzumab-PET-CT scan with standard radiographic imaging for staging patients with gastric cancer.

OUTLINE:

Patients receive copper Cu 64-DOTA-trastuzumab intravenously (IV) on day 1 and then undergo PET/CT scan on days 2 or 3.

After completion of study, patients are followed up for 15 days and periodically for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologic diagnosis of gastric or gastroesophageal junction adenocarcinoma
* Two patients must be HER2 3+ by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH) positive
* Either the primary tumor or at least one of the metastatic lesions must be >= 2 cm
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy of >= 3 months
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of copper Cu 64-DOTA administrations and must have agreed to use an effective contraceptive method; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for four months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* CT/magnetic resonance imaging (MRI) scan must be obtained within 4 weeks prior to study entry
* Patients must have normal cardiac ejection fraction
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* All toxicities should recover to grade 0 or 1 prior to day 1

Exclusion Criteria:

* Impaired cardiac function including any one of the following: complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (< 50 beats per minute), QT interval corrected by Fridericia's formula (QTcF) > 450 msec on screening electrocardiogram (ECG), or right bundle branch block + left anterior hemiblock (bifascicular block)
* Presence of atrial fibrillation
* Previous history of angina pectoris or acute myocardial infarction (MI) within 6 months
* Congestive heart failure (New York Heart Association functional classification III-IV)
* Uncontrolled hypertension (mmHg > 160 systolic or > 90 diastolic)
* Patients should not have active infections or concurrent neoplastic disease except for skin cancer
* Patients may not be receiving any other investigational agents
* At the time of enrollment, patients may not have received any biological, chemotherapy, or radiation therapy
* Patients who may not have received trastuzumab within the prior 6 months for any other reason
* Patients who are pregnant
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanghee Woo, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Copper Cu 64-DOTA-trastuzumab PET Scan): Patients will receive 45 mg trastuzumab over 15 minutes prior to the administration of 64Cu -DOTA-trastuzumab, which includes 5 mg of trastuzumab. Imaging will be performed on a GE Discovery 16 Ste PET-CT scanner (axial field of view 15.4 cm). PET-CT images will be performed in 3D mode (septa retracted) and corrected for tissue attenuation based on co-registered CT acquired during the same examination. PET-CT images will be reconstructed with spatial resolution of approximately 9 mm full-width-at-half maximum using an iterative algorithm. Patients will be injected via a peripheral vein with 15 mCi of 64Cu-DOTA-trastuzumab. PET-CT scanning of 64Cu will be performed between 24 and 48 hours post injection. At 24 hours, the concentration of 64Cu-DOTA-trastuzumab will allow for whole body PET-CT imaging within the same amount of time required to image the abdomen and pelvis at 48 hours due to the half life of the radiotracer. PET-CT images will be compared to standard MRI or CT scans.
Period: Overall Study
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET Scan)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET Scan)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 64 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of HER2 Negative, Positive, or Equivocal Participants With Either Negative or Positive Tumor Readings
Description: The reading of the 64CuDOTA-trastuzumab-PET imaging of the study subjects were performed by two radiologists, one who read the first scan and the second nuclear radiologist read the remaining seven scans. To eliminate potential bias, the second nuclear radiologist was blinded to the HER2 status of the tumors as well as the location of the tumor until radiolabeled uptake was measured. XD (version 3.6; Miranda Medical) was used for image analysis.Tumor visualized as "hot" relative to adjacent tissue reported per radiologist as negative, positive, equivocal or unknown.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET Scan)
Number analyzed (Participants) | 8
participants
  HER2 Negative, Tumor Visual Negative | 5
  HER 2 Positive, Tumor Visual Negative | 1
  HER 2 Equivocal, Tumor Visual Negative | 2
  HER2 Negative, Tumor Visual Positive | 0
  HER 2 Positive, Tumor Visual Positive | 0
  HER 2 Equivocal, Tumor Visual Positive | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 2 years and 4 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET Scan)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Copper Cu 64-DOTA-trastuzumab PET Scan) (N=8)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A total of 8 of the planned 22 gastric adenocarcinoma subjects met eligibility and completed the imaging with 64CuDOTA-Trastuzumab-PET/CT during the 3-year grant period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT01939275/Prot_SAP_001.pdf